CLINICAL TRIAL: NCT04798599
Title: Using Information and Communication Technologies (ICTs) to Solve the Repressed Demand for Primary Dental Care in the SUS Due to the COVID-19 Pandemic
Brief Title: Information and Communication Technologies (ICTS) in Dentistry for SUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of Paraíba (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mariana Minatel Braga, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TeleDent-COVID19
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries in Children; Dental Diseases
Keywords: Child; COVID-19; Information Technology
MeSH Terms: conditions — Stomatognathic Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: This protocol refers to a randomized, patient-controlled study on a waiting list, nested to a before-after type study to be conducted in a cell unit, simulating a basic dental health unit. Next, a modelling study was idealized, prospecting the situation found for the reality and integral demand of the Unified Health System.
  The "before-after" study was designed to measure the positive and negative effects resulting from telecare implementation in primary care for children. The randomised controlled study evaluates the impact of teleservice implementation from the patient´s and parents perception and allows comparison with a reference. For that, children potentially eligible for the study will initially be randomized to one group (intervention vs waiting list). On the waiting list, participants will receive the intervention (standardized telecare) and will be evaluated for outcomes of interest two weeks later.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: One researcher, who will not participate in teleconsultations (intervention), will be responsible for the questionnaires before the intervention and will randomize the patients. This same researcher will distribute the patients randomly among the dentists responsible for teleconsultations. Dentists will also be blind as to the allocation of the patient to the groups. Also, to the patients/families, it will be not mentioned which group participants are part of. An external operator will be responsible for collecting information about the outcome (questionnaire after the interventions) will also not know which group the patient was allocated. As only the researcher responsible for randomization will know which group the patient belongs to and coordinate all operational parts of the teleconsultations, investigators can ensure the other operators and participants' blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention group there will be the application of the intervention - use of telemonitoring and teleorientation applied to children in primary care in Dentistry.
  Interventions: Other: Telemonitoring and teleorientation
- Waiting list (Active Comparator): In the control group, children waiting to be booked to the intervention (in implementation in the unit because of the pandemic) will be evaluated for the outcomes. Only after the evaluation, the control group's children will be invited to perform the teleconsultation (proposed intervention).
  Interventions: Other: Control Group - Waiting list

INTERVENTIONS:
Other: Telemonitoring and teleorientation — Teleservice will be performed through a digital platform (Video for Health" - V4H). The service will consist of: a) recognition of the condition identified in the pandemic period, including updates on medical history, current oral health condition, search for dental care in other units, need for referral, change of hygiene habits, b) realization of diet guidance, hygiene and other necessary habits, made from a situational recognition of such habits, c) targeting the needs presented, in which individualized counselling will be given seeking to meet the demand presented by that family nucleus. A dental form developed on the digital platform Google Forms will serve as a guide for the performance of the service and where the collected data will be formally recorded. The guidelines, although individualized for the needs of each child, will follow a pre-defined and standardized structure and based on the best evidence available in the subject.
  Arms: Intervention
Other: Control Group - Waiting list — No intervention (at least, until the time frame for outcome assessment)
  Arms: Waiting list

SUMMARY:
At the time of the COVID-19 pandemic, thousands of children had their dental care interrupted or postponed, generating a pent-up demand for primary care. In order to minimize the impact of this outage of face-to-face care, information and communication technologies could be an alternative and even likely to be envisioned within the Brazilian Unified Health System (SUS). In this sense, this study sought to show the impact of the use of information and communication technologies (ICT) in the resolution of the pent-up demand for primary dental care to children in the SUS, due to the COVID-19 pandemic, proposing the use of telemonitoring, teleorientation and telescreening to resolve and address demands arising from this outage in primary elective care. The impact of the use of these strategies will be measured in terms of problem-solving, reduction of waiting time to resolve complaints and caregivers' perception about received care. For this, two clinical studies were designed and a primarily trial-based economic evaluation was planned. Mathematical models will be used to transpose these results into the reality of the SUS, in view of the State Health Secretariat of São Paulo and different Brazilian scenarios. Finally, the investigators also aim to study the possibility of implementing these technologies mentioned in the daily life of the SUS, even after a pandemic, and to check the possibility of incorporating and costing them, as well as exploring possible social impact and relationship with possible inequities in health.

DETAILED DESCRIPTION:
Project Objectives:

This proposal has as a general objective to show the impact of the use of information and communication technologies (ICT) on the resolution of the pent-up demand for primary dental care to children in the SUS, due to the COVID-19 pandemic.

To this do so, the following specific objectives are defined:

1. To identify the pent-up demand for the outage of dental care and the benefits and difficulties, as well as the perception of users, in the implementation of new strategies of non-face-to-face care based on technology (teleservice), using a primary care cell unit for children and prospecting, through models, this situation for the scenario of the Unified Health System (SUS).
2. Perform different forms of economic evaluation to measure whether the gains achieved with the implementation of teleservice (telescreening, teleorientation and telemonitoring) compensate for the additional costs possibly associated with it, or whether teleservice modalities are associated with long-term resource savings, taking into account the implementation sized for the Brazilian public health system.
3. Explore how the introduction of these technologies could benefit the SUS in the trans and post-pandemic period, contribute to the correction of possible inequities in health care and other social aspects, as well as result in possible differences when different Brazilian scenarios are explored.

ELIGIBILITY:
Inclusion Criteria:

- Children from 3 to 13 years old who are involved in clinical studies and who already undergo follow-up from 6 to 60 months in the mobile dental unit.

Exclusion Criteria:

* Guardian´s participants) who do not accept to participate in the research and if participants accept.
* Children who do not assent with participation in the research (when already literate). - For children aged 3 to 6 years, included in the research, the waiver of the need to fill out the term of free and informed assent was requested, considering that these children are not literate and would not be able to write, to assent with the participation. t

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 368 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Family/patient´s perception about the dental care | 2 weeks after intervention (or one week of waiting - in the case of the control group)
  Evaluation of the quality of dental care to be measured by the SERVQUAL questionnaire (a multi-dimensional research instrument) - total of 22 items and 5 dimensions, comprising 4 items to capture tangibles, 5 items to capture reliability, 4 items for responsiveness, 4 items for assurance and 5 items to capture empathy.
  A total of 100 points is allocated among the five dimensions. The participants evaluate the degree to which they perceived the proposed service. To identify participants' perceptions, one item asked, "How do you feel about these service attributes that are already provided?", which was scored on a 5-point Likert-type scale of "very bad (1)" to "very good (5)."

SECONDARY OUTCOMES:
Increment in caries experience since the interruption of dental care | 1 year after intervention
  Clinical examination focused using dmft and DMFT indices and comparison to those. An previously recorded in participant´s records, resulting in the difference between the indices between these moments (DMFT+dmft final - DMFT+dmft when treatment was interrupted). An examiner unaware of baseline conditions will assess these indices.
Increment or changes in the needs for dental treatment | 1 year after intervention
  Clinical examination focused in detecting if there is need for dental treatment or not (including untreated caries, need for restoration repair, need of gingival or periodontal treatment, need for extractions for any reason). An examiner unware of baseline conditions will assess such needs.
Demand resolution after intervention | 2 weeks after intervention
  Interview for checking about the resolution of demands pointed out during the baseline consultation.
Need for reorientation about oral hygiene | 2 weeks, 3 months, 6 months, 1 year after intervention
  Interview for checking doubts about oral hygiene and checklist of items to be accomplished during oral hygiene demonstrated by child. An external examiner will evaluate all listed items. In case of any one is not checked, the need of reorientation is considered.
Perception of caregivers regarding primary care and dental care. | 2 weeks after intervention
  Semi-structured interviews, applied with guided questions to try to assess participants' and parents' perception, as well as potential barriers and facilitators associated with dental care during the pandemic period with the caregivers of the children who followed the teleservice. For this, individual interviews will be recorded and transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, PhD, Principal Investigator — USP
Locations (1):
- University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natal KH, Machado TG, Bracco F, Lemos LI, Vigano ME, Machado GM, Yampa-Vargas JD, Raggio DP, Mendes FM, Imparato JCP, Lucena EHG, Cavalcanti YW, Silva CI, Souza Filho GL, Macedo MCS, Carrer FCA, Braga MM. Using information and communication technologies (ICTs) to solve the repressed demand for primary dental care in the Brazilian Unified Health System due to the COVID-19 pandemic: a randomized controlled study protocol nested with a before-and-after study including economic analysis. BMC Oral Health. 2022 Apr 7;22(1):112. doi: 10.1186/s12903-022-02101-9. PMID 35392886